CLINICAL TRIAL: NCT07273604
Title: Psychological Intervention in Multiple Sclerosis: Efficacy in the Treatment of Anxiety-depressive Symptoms and Cognitive Impairment.
Brief Title: Psychological Interventions for Multiple Sclerosis: Effects on Anxiety, Depression, and Cognition.
Acronym: MS-PSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moisés Bermúdez Hernández (Other)
Collaborators: University of La Laguna (Other)
Responsible Party: Sponsor-Investigator, Moisés Bermúdez Hernández, Principal Investigator and Researcher, Hospital Universitario Nuestra Señora de Candelaria (HUNSC); Professor of Psychology, University of La Laguna, University of La Laguna
Organization: University of La Laguna (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUNSC_ULL_MS_PSY2015; PI-60/14 (Other: Universidad de La Laguna (ULL) and Hospital Universitario Nuestra Señora de Candelaria (HUNSC))
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting; Anxiety; Depression; Cognitive Impairment; Emotional Well-being; Cognitive Behavior Therapy
Keywords: Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Cognitive Behavioral Therapy; Psychophysiological Regulation Therapy; Anxiety; Depression; Cognitive Impairment; Emotional Well-being; Quality of Life; Fatigue; Randomized Controlled Trial; Psychological Intervention
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Anxiety Disorders; Depression; Cognitive Dysfunction; Multiple Sclerosis; Fatigue | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study employed a three-arm randomized controlled design with participants allocated to Cognitive Behavioral Therapy (CBT), Psychophysiological Regulation Therapy (PRT), or Standard Care (waiting list). Interventions were group-based over 12 weekly sessions, with assessments at baseline and post-intervention. Both CBT and PRT followed structured programs aimed at improving stress coping and reducing anxiety-depressive symptoms through psychoeducation, mindfulness, and psychophysiological regulation. Sessions combined didactic content, group exercises, and homework. CBT emphasized behavioral activation, cognitive restructuring, self-instruction, and social skills training, whereas PRT focused on psychophysiological self-regulation, relaxation, breathing control, and biofeedback exercises.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to participants' group allocation. Participants and therapists were aware of the assigned intervention, but evaluators conducting clinical and neuropsychological assessments did not have access to treatment information to minimize bias in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Therapy (CBT) (Experimental): Participants receive a structured 12-week cognitive-behavioral group intervention designed to improve stress coping and reduce anxiety-depressive symptoms. The program includes psychoeducation, mindfulness, behavioral activation, cognitive restructuring, self-instruction training, and social skills development.
  Intervention: Behavioral: Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Psychophysiological Regulation Therapy (PRT) (Experimental): Participants receive a structured 12-week group intervention emphasizing psychophysiological self-regulation. The program includes psychoeducation, mindfulness, relaxation, breathing control, and biofeedback-based exercises aimed at reducing emotional distress and enhancing self-regulation.
  Interventions: Behavioral: Psychophysiological Regulation Therapy (PRT)
- Standard Care (SC) (No Intervention): Participants in the control group remain on a waiting list and receive standard medical care provided by the Multiple Sclerosis Unit during the study period. After study completion, they are offered participation in one of the active interventions.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — A structured 12-week group-based cognitive-behavioral intervention including psychoeducation, mindfulness training, behavioral activation, cognitive restructuring, self-instruction training, and social skills development. Designed to improve coping, reduce anxiety-depressive symptoms, and enhance cognitive and emotional functioning.
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: Psychophysiological Regulation Therapy (PRT) — A structured 12-week group-based intervention emphasizing psychophysiological self-regulation through psychoeducation, mindfulness, relaxation, breathing control, and biofeedback-based exercises to reduce emotional distress and promote physiological balance.
  Arms: Psychophysiological Regulation Therapy (PRT)

SUMMARY:
This study evaluated the efficacy of two structured psychological interventions for patients with relapsing-remitting multiple sclerosis (RRMS). The main goal was to determine whether a Cognitive Behavioral Therapy (CBT)-based program and a Psychophysiological Regulation Therapy (PRT) improved emotional well-being and cognitive functioning compared with Standard Care (SC).

A total of 140 participants with mild to moderate disability and disease duration between 5.5 and 8.5 years were randomly assigned to one of three groups: CBT, PRT, or SC (waiting list). Each intervention was delivered in small groups over 12 weekly sessions. Assessments were conducted before and after treatment using validated clinical and neuropsychological measures.

Results were analyzed to explore the effectiveness of both interventions in reducing anxiety and depressive symptoms and enhancing cognitive performance. The study aimed to provide evidence for the inclusion of psychological therapies as complementary treatments in comprehensive care for multiple sclerosis patients.

DETAILED DESCRIPTION:
A randomized controlled trial design will be conducted with allocation to the following groups: treatment group (cognitive-behavioral intervention group, psychophysiological reduction - low performance - and neuropsychological rehabilitation) or control group (waiting list). Assessments will be carried out before and immediately after treatment, and at a six-month follow-up after therapy completion. Additionally, a follow-up magnetic resonance imaging (MRI) will be performed after the intervention, within a period of 1 to 3 months, and again at 6 months post-treatment. This neuroimaging activity is included as part of the clinical practice of the Multiple Sclerosis Unit. Participants: A total of 140 patients with clinically defined relapsing-remitting Multiple Sclerosis (MS) will be studied. Inclusion criteria will include minimal to mild disability according to the Expanded Disability Status Scale (EDSS) (EDSS: 0-3.5), mild to moderate cognitive impairment (BRB-N: up to two subtests with scores <2 SD), and presence of anxiety and/or depressive symptoms (HADS: scores >8 on one or both subscales; BDI-II: scores >8). Participants will be recruited from the Multiple Sclerosis Unit of the University Hospital Nuestra Señora de Candelaria (HUNSC) in Santa Cruz de Tenerife. The sample size calculation was based on the assumption that, to achieve a 90% power for detecting effects on primary measures (BDI-II, HADS, ISRA, BRB-N, etc.). The sample size was calculated based on an ANOVA design (medium effect size, d = 0.5; α = 0.05; power = 80%), estimating a required total of 156 participants (52 per group).

. This estimate may be adjusted throughout data collection due to variability in measures specific to this population. Experience with the initial participant groups and their resulting data will allow refinement of these estimates. Evidence highlights that people with MS exhibit unusually low levels of help-seeking behavior for anxiety and depressive symptoms, emphasizing the need for systematic screening. The Multiple Sclerosis Unit currently follows 587 diagnosed patients. This study also aims, based on initial findings, to broaden inclusion criteria according to preliminary results and to establish comparisons among different forms of MS, thereby improving the external validity of the study. This approach is grounded in the reflections of several authors who note that overly restrictive inclusion criteria (e.g., symptoms, comorbidities) may limit the generalizability of clinical trial results to routine clinical practice. They propose ensuring adequate representation of problems, settings, and therapies, along with systematic treatment monitoring and flexibility in interventions-while maintaining detailed information on their active components. Procedure and Timeline Pre-treatment Evaluation Neurological Evaluation: Initial selection of patients will be conducted at the Multiple Sclerosis Unit of the Neurology Service at the University Hospital Nuestra Señora de Candelaria. A standardized neurological protocol will be requested, including the most relevant clinical history data and neurological examination results. Clinical inclusion criteria: clinically defined relapsingremitting MS and minimal to mild disability level. Psychological Evaluation: Among patients meeting clinical inclusion criteria, an interview will be conducted to identify those reporting cognitive and emotional complaints (including an interview with relatives). Motivation and willingness to collaborate will also be assessed. Upon obtaining informed consent, the evaluation protocol will be administered to determine fulfillment of cognitive and emotional inclusion criteria. Patients meeting the criteria will be randomly assigned to either the intervention group or the control group (waiting list without intervention), considering their anxiety and depression scores as well as cognitive impairment levels. The inclusion period will last approximately four months. Treatment Phase Patients in the treatment group will complete the psychological intervention program over 12 weeks (one weekly session lasting 1 hour and 30 minutes), plus two follow-up sessions. The intervention will follow a cognitive-behavioral framework and consist of a specific program tailored to the characteristics of the identified deficits. It will include didactic sessions, group discussions, and practical exercises. Post-treatment Evaluation This will take place during the week following the end of treatment and will include: Neurological Evaluation: assessment of disability level (EDSS).

Psychological Evaluation: assessment of cognitive, emotional, and quality-of-life variables. Follow-up Evaluation A follow-up assessment will be carried out six months after treatment completion, applying the same evaluation protocol as in previous phases.

The control group will be evaluated at the same time points as the intervention group.

All phases of the study will be conducted at the Multiple Sclerosis Unit of the University Hospital Nuestra Señora de Candelaria (HUNSC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting multiple sclerosis according to standard clinical criteria.
* Expanded Disability Status Scale (EDSS) score between 0 and 3.5.
* Mild to moderate cognitive impairment defined as: up to two BRB-N subtests with scores < -2 SD.
* Presence of anxiety or depressive symptoms defined as:
* HADS: score > 8 on one or both subscales, and/or
* BDI-II: score > 8.
* Stable disease-modifying treatment for ≥ 3 months.
* Ability to provide written informed consent.

Exclusion Criteria:

* Progressive forms of multiple sclerosis (SPMS or PPMS).
* Severe cognitive impairment preventing participation in psychological sessions.
* Active psychiatric or neurological disorders unrelated to MS.
* Participation in another psychological or pharmacological intervention study.
* Recent initiation or modification of disease-modifying treatment (< 3 months).
* Substance abuse or dependence within the past year.
* Inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale (FSS) - Total Score | Baseline and 12 weeks.
  Description: Change in fatigue severity measured with the Fatigue Severity Scale (FSS; Krupp et al., 1989).
  Scale range: 9-63 points (9 items scored 1-7). Interpretation: Higher scores indicate greater fatigue severity.
Multiple Sclerosis Quality of Life-54 (MSQoL-54) - Total and Subscale Scores | Baseline and 12 weeks.
  Description: Change in quality of life measured with the Multiple Sclerosis Quality of Life-54 (MSQoL-54; Vickrey, Hays, Harooni, Myers & Ellison, 1995), including physical and mental health composite scores and individual subscales.
  Scale range: 0-100 points. Interpretation: Higher scores indicate better quality of life.
Multiple Sclerosis Neuropsychological Questionnaire (MSNQ) - Total Score | Baseline and 12 weeks.
  Description: Change in perceived cognitive functioning measured with the Multiple Sclerosis Neuropsychological Questionnaire (MSNQ; Benedict et al., 2003).
  Scale range: 0-60 points. Interpretation: Higher scores indicate greater perceived cognitive impairment.
Verbal Selective Reminding Test (SRT) - Total Recall Score | Baseline and 12 weeks.
  Change in verbal learning and memory performance measured with the Verbal Selective Reminding Test (SRT), part of the BRB-N (Rao, 1990). (Scale range 0-72). Interpretation: Higher scores indicate better performance.
10/36 Spatial Recall Test (SPART) - Total Recall Score | Baseline and 12 weeks.
  Description: Change in visuospatial learning and memory measured with the 10/36 Spatial Recall Test (SPART), part of the BRB-N (Rao, 1990).
  Scale range: 0-36. Interpretation: Higher scores indicate better performance.
Paced Auditory Serial Addition Test (PASAT) - 3-Second Version | Baseline and 12 weeks.
  Description: Change in complex attention and working memory measured with the PASAT (3-second version), part of the BRB-N (Rao, 1990).
  Scale range: 0-60 correct responses. Interpretation: Higher scores indicate better performance.
Symbol Digit Modalities Test (SDMT) - Oral Version | Baseline and 12 weeks.
  Description: Change in attention and processing speed measured with the Symbol Digit Modalities Test (SDMT), part of the BRB-N (Rao, 1990).
  Scale range: 0-110 correct responses. Interpretation: Higher scores indicate better performance.
Controlled Oral Word Association Test (COWAT) - Semantic Fluency ("Animals" Category) | Baseline and 12 weeks.
  Description: Change in semantic verbal fluency measured with the Controlled Oral Word Association Test (COWAT), Semantic Fluency subtest (animals category).
  Scale range: Number of correct animals named in 60 seconds (typically 0-40). Interpretation: Higher scores indicate better performance.
Controlled Oral Word Association Test (COWAT) - Phonemic Fluency (F-A-S Letters) | Baseline and 12 weeks.
  Description: Change in phonemic verbal fluency measured with the Controlled Oral Word Association Test (COWAT), Phonemic Fluency subtest (letters F, A, and S).
  Scale range: Total number of correct words generated across the three letters in 60 seconds each (typically 0-60).
  Interpretation: Higher scores indicate better performance.
Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A) | Baseline and 12 weeks.
  Description: Change in anxiety symptoms measured with the Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A; Zigmond & Snaith, 1983).
  Scale range: 0-21 points. Interpretation: Higher scores indicate greater anxiety severity.
Beck Depression Inventory-II (BDI-II) - Total Score | Baseline and 12 weeks.
  Description: Change in depressive symptoms measured with the Beck Depression Inventory-II (BDI-II; Beck et al., 1996).
  Scale range: 0-63 points. Interpretation: Higher scores indicate greater depressive severity.
Inventario de Situaciones y Respuestas de Ansiedad (ISRA) - Total Score | Baseline and 12 weeks.
  Description: Change in cognitive, physiological, and motor anxiety responses measured with the Inventario de Situaciones y Respuestas de Ansiedad (ISRA; Miguel-Tobal & Cano-Vindel, 1994).
  Scale range: 0-100+ (higher scores = greater anxiety response). Interpretation: Higher scores indicate greater anxiety reactivity.

SECONDARY OUTCOMES:
Recent Life Changes Questionnaire (RLCQ) - Total Score | Baseline and 12 weeks.
  Description: Change in perceived stress measured with the Recent Life Changes Questionnaire (RLCQ; Holmes & Rahe, 1967; Spanish adaptation: González & Morera, 1983).
  Scale range: 0 to 100+ life change units (LCUs), depending on the number and weight of events endorsed.
  Interpretation: Higher scores indicate greater perceived stress and higher adjustment demand.
Symptom Checklist-90-Revised (SCL-90-R) - Global Severity Index (GSI) | Baseline and 12 weeks.
  Description: Change in general psychopathological symptoms measured with the Symptom Checklist-90-Revised (SCL-90-R; Derogatis, 1994), using the Global Severity Index (GSI).
  Scale range: 0-4 (mean item score across 90 items rated 0 to 4). Interpretation: Higher scores indicate greater psychopathological symptom severity.
Cognitive Triad Inventory (CTI) - Total Score | Baseline and 12 weeks.
  Description: Change in depressive cognitive schemas measured with the Cognitive Triad Inventory (CTI; Beckham et al., 1986).
  Scale range: 36-252 points (36 items scored 1-7). Interpretation: Higher scores indicate more negative/depressive cognitive schemas about self, world, and future.
Intolerance of Uncertainty Scale (IUS) - Total Score | Baseline and 12 weeks.
  Description: Change in intolerance of uncertainty measured with the Intolerance of Uncertainty Scale (IUS; Freeston et al., 1994).
  Scale range: 27-135 points (27 items scored 1-5). Interpretation: Higher scores indicate greater intolerance of uncertainty.
Social Support Questionnaire (SSQ-6) - Total Score | Baseline and 12 weeks.
  Description: Change in perceived social support measured with the Social Support Questionnaire (SSQ; Sarason et al., 1983).
  Scale range: Typically 0-9 for the number of supports (SSQ-6) and 1-6 for satisfaction (SSQ-S), depending on the scoring method used.
  Interpretation: Higher scores indicate greater perceived social support (more available supports and/or higher satisfaction).
Pittsburgh Sleep Quality Index (PSQI) - Total Score | Baseline and 12 weeks.
  Description: Change in sleep quality measured with the Pittsburgh Sleep Quality Index (PSQI).
  Scale range: 0-21 points. Interpretation: Higher scores indicate worse sleep quality.
MRI Lesion Activity and Lesion Load | Baseline and 12 weeks.
  Change in brain lesion activity (number of new/enlarging T2 lesions and gadolinium-enhancing lesions) and total lesion load (total T2 lesion volume) obtained from routine clinical magnetic resonance imaging (MRI) scans.
Duke-UNC Functional Social Support Questionnaire (DUFSS) - Total Score | Baseline and 12 weeks
  Description: Change in functional social support measured with the Duke-UNC Functional Social Support Questionnaire (DUFSS; Broadhead et al., 1988; Spanish validation by Bellón et al., 1996).
  Scale range: 5-55 points (11 items scored 1-5). Interpretation: Higher scores indicate greater functional social support.

OTHER OUTCOMES:
Disease-Modifying and Symptomatic Treatment Status | Baseline and 12 weeks.
  Changes in disease-modifying therapies (DMTs) and symptomatic treatments recorded at each assessment point. Includes initiation, discontinuation, or dose adjustments of any MS-related medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology, University of La Laguna Department of Clinical Psychology, Psychobiology and Methodology of Behavioral Sciences Campus de Guajara, Calle Heraclio Sánchez, s/n 38200 San Cristóbal de La Laguna, Santa Cruz de Tenerife Spain, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available upon reasonable request to the corresponding author, Dr. Moisés Bermúdez Hernández (mbermudh@ull.edu.es), for academic and non-commercial research purposes. Data will be fully anonymized in compliance with institutional and ethical regulations and the European General Data Protection Regulation (GDPR).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting documents will be available beginning 12 months after publication of the main results and will remain accessible for 5 years thereafter.
Access Criteria: Qualified researchers affiliated with academic or non-profit institutions may request access to de-identified individual participant data (IPD) and supporting documents (protocol, SAP, ICF, CSR) for scientific and non-commercial purposes. Requests must be submitted to the corresponding author, Dr. Moisés Bermúdez Hernández (mbermudh@ull.edu.es). Access will be granted following review and approval by the study's ethics committee and in compliance with GDPR and institutional data-sharing policies.

REFERENCES:
- [Background] Scandiffio J, Langer LK, Senthilnathan V, Feng G, Sureshkumar A, Bromberg M, Babineau J, Donkers SJ, Knox KB, Bruno T, Walker LAS, Bayley MT, Simpson R. Effects of psychological therapies in people with multiple sclerosis: a systematic review and network meta-analysis of randomized controlled trials. J Neurol. 2025 Aug 20;272(9):584. doi: 10.1007/s00415-025-13315-6. PMID 40833620
- [Background] Lucien A, Francis H, Wu W, Woldhuis T, Gandy M. The efficacy of cognitive behavioural therapy for depression and anxiety in multiple sclerosis: A systematic review and meta-analysis. Mult Scler Relat Disord. 2024 Nov;91:105858. doi: 10.1016/j.msard.2024.105858. Epub 2024 Sep 3. PMID 39276596
- [Background] Moss-Morris R, McCrone P, Yardley L, van Kessel K, Wills G, Dennison L. A pilot randomised controlled trial of an Internet-based cognitive behavioural therapy self-management programme (MS Invigor8) for multiple sclerosis fatigue. Behav Res Ther. 2012 Jun;50(6):415-21. doi: 10.1016/j.brat.2012.03.001. Epub 2012 Mar 13. PMID 22516321
- [Background] De Meo E, Portaccio E, Bonacchi R, Giovannoli J, Niccolai C, Amato MP. An update on the treatment and management of cognitive dysfunction in patients with multiple sclerosis. Expert Rev Neurother. 2025 Feb;25(2):227-243. doi: 10.1080/14737175.2025.2450788. Epub 2025 Jan 16. PMID 39801437
- [Background] Cuijpers P, Karyotaki E, Weitz E, Andersson G, Hollon SD, van Straten A. The effects of psychotherapies for major depression in adults on remission, recovery and improvement: a meta-analysis. J Affect Disord. 2014 Apr;159:118-26. doi: 10.1016/j.jad.2014.02.026. Epub 2014 Feb 24. PMID 24679399
- [Background] Amato MP, Langdon D, Montalban X, Benedict RH, DeLuca J, Krupp LB, Thompson AJ, Comi G. Treatment of cognitive impairment in multiple sclerosis: position paper. J Neurol. 2013 Jun;260(6):1452-68. doi: 10.1007/s00415-012-6678-0. Epub 2012 Nov 23. PMID 23180174